CLINICAL TRIAL: NCT04688333
Title: E-Interventions to Treat Fear of Cancer Recurrence for Patients With Localized Renal Cell Carcinoma
Brief Title: iConquerFear Program for the Treatment of Fear of Cancer Recurrence in Patients With Localized Renal Cell Carcinoma
Status: Withdrawn | Type: Observational
Why Stopped: Feasibility
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20133; NCI-2020-04378 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20133 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-09-10; First posted 2020-12-30 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Supportive care (iConquerFear program, questionnaires): Patients complete 5 sessions of iConquerFear program online over 5 weeks. Patients also complete questionnaires at baseline, after the intervention, and 2 months later.
  Interventions: Other: Internet-Based Intervention - Complete iConquerFear program; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention - Complete iConquerFear program — Online adaptation of a highly effective face-to-face treatment for fear of recurrence.
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This trial investigates whether an online intervention, iConquerFear, can reduce fear of cancer coming back (recurrence) and anxiety in patients with renal cell carcinoma that is restricted to the site of origin, without evidence of spread (localized). This intervention is an online adaptation of a highly effective face-to-face treatment for fear of recurrence that teaches strategies for: controlling worry and excessive threat monitoring, modifying unhelpful beliefs about worry, developing appropriate monitoring and screening behaviors, addressing cancer-related existential change, promoting values-based goal setting, and reducing uncertainty by providing information about cancer and treatment. The information learned may help others with renal cell carcinoma who also have a fear of cancer recurrence.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess feasibility and acceptability of the iConquerFear program for patients with renal cell carcinoma (RCC).

II. To assess preliminary effects of the program on Fear of Cancer Recurrence-7 item scale (FCR-7), Patient-Reported Outcomes Measurement Information System (PROMIS)-anxiety, PROMIS-depression, and Functional Assessment of Chronic Illness Therapy-General (FACT-G).

III. Explore differences in feasibility and efficacy of iConquerFear by sociodemographic or clinical factors.

OUTLINE:

Patients complete 5 sessions of iConquerFear program online over 5 weeks. Patients also complete questionnaires at baseline, after the intervention, and 2 months later.

ELIGIBILITY:
Inclusion Criteria:

* Sufficiently fluent in English
* Cytologically or pathologically verified diagnosis of RCC
* Undergone nephrectomy with negative margins (NOTE: Patients with other local definitive therapies, e.g., radiofrequency ablation or stereotactic ablative radiotherapy [SABR], would not be candidates for this protocol)
* No evidence of metastatic disease (including at a minimum computed tomography [CT] of the chest, abdomen and pelvis for staging)
* Internet access and basic computer skills
* Moderate to severe fear of cancer recurrence (FCR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal Cell Carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2023-08-27 (Estimated); Study Completion 2023-08-27 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Accrual | 1 year
  at least 90% of the desired accrual goal is reached within 12 months
Feasibility - completion of Interventions | 1 year
  At least 70% of patients complete 3/5 intervention sessions, assessed as follows:
  i. ≥70% of patients complete first intervention session ii. ≥70% of patients complete second intervention session iii. ≥70% of patients complete third intervention session
Feasibility - retention/evaluation | 1 year
  ≥70% of patients have at least 2 of 3 evaluable time points, assessed as follows: i. All patients will have timepoint 1 assessment, which is required at time of accession ii. ≥70% of patients must be evaluable at timepoint 2 or timepoint 3 [in rare cases, patients will skip in intermediary time point but compelete a later timepoint evaluation]

SECONDARY OUTCOMES:
Preliminary effects of iConquerFear program - FCR 7 | Baseline (T1), immediately after the intervention expected at 5 weeks after baseline (T2), and at 2 months follow-up (T3, 2 months following T2)]
  Analysis of Variance (ANOVA) will be used to explore changes in scores over time, separately for the metrics obtained from Fear of Cancer Recurrence-7 item scale (FCR-7)
  All instruments will be scored according to validated instructions. All available time points will be used in each analysis.
  Fear of Cancer Recurrence-7. This is a 7-item scale that assesses the degree of FCR, with a cutoff score of 17 or above indicative of moderate and a cutoff score of 27 or above indicative of severe FCR.
Preliminary effects of iConquerFear program - (PROMIS)-Anxiety | Baseline (T1), immediately after the intervention expected at 5 weeks after baseline (T2), and at 2 months follow-up (T3, 2 months following T2)]
  Analysis of Variance (ANOVA) will be used to explore changes in scores over time, separately for the metrics obtained from Patient-Reported Outcome Measurement Information System (PROMIS)-Anxiety.
  All instruments will be scored according to validated instructions. All available time points will be used in each analysis.
  PROMIS Emotional Distress: Anxiety. This 8-item measure assesses symptoms of anxiety on a 5-point scale (1=never, 5=always). Scores range from 7-35 with higher scores indicating greater severity of anxiety.
Preliminary effects of iConquerFear program - PROMIS -depression | Baseline (T1), immediately after the intervention expected at 5 weeks after baseline (T2), and at 2 months follow-up (T3, 2 months following T2)]
  Analysis of Variance (ANOVA) will be used to explore changes in scores over time, separately for the metrics obtained from Patient-Reported Outcome Measurement Information System (PROMIS)-depression.
  All instruments will be scored according to validated instructions. All available time points will be used in each analysis.
  PROMIS Emotional Distress: Depression. This 8-item measure assesses symptoms of depression on a 5-point scale (1=never, 5=always). Scores range from 8-40 with higher scores indicating greater severity of depression.
Preliminary effects of iConquerFear program - FACT-G | Baseline (T1), immediately after the intervention expected at 5 weeks after baseline (T2), and at 2 months follow-up (T3, 2 months following T2)]
  Analysis of Variance (ANOVA) will be used to explore changes in scores over time, separately for the metrics obtained from Functional Assessment of Chronic Illness Therapy-General (FACT-G).
  All instruments will be scored according to validated instructions. All available time points will be used in each analysis.
  Functional Assessment of Chronic Illness Therapy-General (FACT-G). A 27-item self-related scale measure QoL across four domains of 'well-being' (physical, social/family, emotional and functional) on a 4-point Likert scale. Scores range from 0-28 for the physical, social/family and functional subscales, 0-24 for the emotional subscale and 0-108 for the total score. Higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — City of Hope Medical Center